CLINICAL TRIAL: NCT01304901
Title: Phase 4 Study of Single Dose of Oral Montelukast When Adding to Standard Treatment in Acute Moderate to Severe Wheezing in Preschool Children.
Brief Title: Effect of Addition of Single Dose of Oral Montelukast to Standard Treatment in Acute Asthma in Preschool Children.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kecioren Education and Training Hospital (Other)
Responsible Party: Principal Investigator, Cem Hasan Razi, MD, Kecioren Education and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B.10.0.İEG-0.15-00-01/5181
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Last update posted 2011-12-20 (Estimated); Status verified 2011-12

CONDITIONS: Asthma; Acute Asthma
Keywords: Acute asthma; Children; Montelukast; Emergency room
MeSH Terms: conditions — Asthma; Emergencies | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1-Montelukast (Active Comparator): Children had received single dose of 4 mg oral montelukast after first dose of nebulized salbutamol and systemic glucocorticoids.
  Interventions: Drug: montelukast 4 mg granule
- 2- Placebo (Placebo Comparator): Children had received single dose of oral placebo montelukast granule after first dose of nebulized salbutamol and systemic glucocorticoids.
  Interventions: Drug: Montelukast placebo granüle

INTERVENTIONS:
Drug: montelukast 4 mg granule — Children had received single dose of 4 mg oral montelukast after first dose of nebulized salbutamol and systemic glucocorticoids.
  Arms: 1-Montelukast
Drug: Montelukast placebo granüle — Children had received single dose of oral placebo montelukast granule after first dose of nebulized salbutamol and systemic glucocorticoids.
  Other Names: Montelukast placebo granule
  Arms: 2- Placebo

SUMMARY:
The purpose of this study is to determine if adding single dose of oral montelukast to the standard treatment of systemic glucocorticoids plus short acting beta-2 agonist for treatment of acute wheezing provide additional clinical benefit in the emergency room.

DETAILED DESCRIPTION:
Systemic corticosteroids and short acting beta-2 agonists are the mainstay treatment of acute asthma, however, little data exists regarding use of leukotriene antagonists in acute asthma. A few studies in adults have shown that oral montelukast also improved pulmonary function when being added to the standard treatment. But in school-age children this clinical benefit could not be demonstrated by adding montelukast to the standard treatment of acute asthma in emergency room. Moreover in preschool children there are no studies on this topic.

The investigators hypothesized that addition of single dose of oral montelukast to standard therapy in acute moderate to severe wheezing may provide additional benefit in the meaning of improvement of pulmonary score and/or proportion of discharge from emergency department in preschool-age children.

ELIGIBILITY:
Inclusion Criteria:

* 6 months to 6 years of age
* With at least three episodes of wheezing in the previous 12 months
* Who presented to the ED with a moderate to severe wheezing episode (defined as a Pulmonary Index Score [PIS] of 7 to 13

Exclusion Criteria:

* Patients who were receiving more than 400 mcg of inhaled budesonide or equivalent per day
* Who had any change in their dose of ICSs in the past 2 months
* Who had taken systemic corticosteroid within 1 months
* Patients who have concurrent pneumonia, croup or suspected foreign body aspiration, a history of cystic fibrosis, bronchopulmonary dysplasia, bronchiolitis obliterans, congenital heart disease, liver or renal disease,sickle cell anemia or immune deficiency were excluded.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Difference of pulmonary index score from baseline to 120 minutes. | 0 to 120 minutes
  İmprovment of pulmonary index score from 0 to 120 minutes was compared bwtween the montelukast and placebo groups.

SECONDARY OUTCOMES:
Proportion of discharge from emergency department. | 120, 180 and 240. minutes
  Proportion of subjects who were discharged from emergency department at 120,180 and 240. minutes were compared between the montelukast and placebo groups.

CONTACTS AND LOCATIONS:
Overall Officials: CEM H RAZİ, M.D., Study Director — Kecioren Education and Training Hospital; ELİF YAĞLI ÇOLAKOĞLU, M.D., Principal Investigator — Kecioren Education and Training Hospital
Locations (1):
- Kecioren Education and Training Hospital, Ankara, Keçiören, Turkey (Türkiye)